CLINICAL TRIAL: NCT03490006
Title: Ultrasound-guided Thoracic Paravertebral Block Versus Ultrasound-guided Thoracic Erector Spinae Plane Block for Pain Management After Unilateral Total Mastectomy: a Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Paravertebral Block in Mastectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient resources to complete study requirements
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, John Alexander, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 012018-081
Record Dates: First submitted 2018-03-20; First posted 2018-04-06 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Pain
Keywords: regional anesthesia; postoperative pain; mastectomy; erector spinae plane block; paravertebral block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two parallel arms. One group will receive erector spinae plane block, and the other will receive paravertebral block.
Who Masked: Outcomes Assessor
Masking Description: The practitioner must know which block to perform, and the patient will be able to deduce which block was performed because paravertebral requires two injections, and erector spinae requires only one injection. The outcomes assessor will not know which group each patient is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paravertebral Block (Active Comparator): For this arm, the initial level will be at T3-4 and an out-of-plane technique to guide the needle tip to a point between the costotransverse ligament and the parietal pleura between the visualized transverse processes. Then, a few milliliters of 0.5% ropivacaine will be injected slowly to displace the pleura ventrally as the paravertebral space fills with local anesthetic. After negative aspiration, the rest of 0.5% ropivacaine (total 10 ml) will be injected in 5 ml increments to further fill the paravertebral space. The procedure will then be repeated in the same exact fashion at the T5-6 level. We will observe local anesthetic spread under real-time ultrasound imaging.
  Interventions: Procedure: Paravertebral Block
- Erector Spinae Plane Block (Experimental): For this arm, the needle tip will be directed under ultrasound guidance using an in-plane technique towards the T5 transverse process until the needle tip contacts os. Then, a few milliliters of ropivacaine will be injected slowly to separate the plane between the erector spinae muscle and the transverse process. After negative aspiration, the rest of the 0.5% ropivacaine will be injected (total 20ml)
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — A relatively recent alternative to the paravertebral block is the thoracic erector spinae plane block, which involves the ultrasound-guided injection of local anesthetic into the interfascial plane deep to the erector spinae muscle at the level of the transverse process. It results in a loss of somatic sensory sensation across multiple unilateral dermatomes due to local anesthetic mediated blockade of the dorsal and ventral rami of the spinal nerve roots. It is increasingly being used due to ease of placing the block and a perception of greater safety. It has been shown to provide pain relief from rib fractures, thoracotomy, and chronic neuropathic pain of the chest wall. However, to date, erector spinae plane block has not been compared with paravertebral block in regards to analgesia with mastectomy surgery, which has been extensively studied.
  Arms: Erector Spinae Plane Block
Procedure: Paravertebral Block — Paravertebral block is a classic regional anesthesia technique that has been in use for over 100 years. It is performed by the injection of local anesthetic into the space between the costotransverse ligament and parietal pleura resulting in blockade of ipsilateral intercostal nerves. It results in a loss of somatic sensation over multiple unilateral dermatomes.
  Arms: Paravertebral Block

SUMMARY:
In this randomized, controlled, observer-blinded study the investigators plan to evaluate ultrasound-guided thoracic paravertebral block (TPVB) and ultrasound-guided thoracic erector spinae plane (TESP) block for postoperative pain management after unilateral total mastectomy without immediate reconstruction.

DETAILED DESCRIPTION:
Despite substantial advances in our understanding of the pathophysiology of pain and availability of newer analgesic techniques postoperative pain is not always effectively treated. Optimal pain management technique balances pain relief with concerns about safety and adverse effects associated with analgesic techniques. Currently, postoperative pain is commonly treated with systemic opioids, which are associated with numerous adverse effects including nausea and vomiting, dizziness, drowsiness, pruritus, urinary retention, and respiratory depression. Use of regional and local anesthesia has been shown to reduce opioid requirements and opioid-related side effects. Therefore, their use has been emphasized. The advent of ultrasound guided regional anesthesia has brought more precision to these techniques, including the ability to visualize the anatomy, perform real-time navigation, and direct observation of local anesthetic spread, as it allows a greater degree of sensory and motor blockade. Thoracic paravertebral block (TPVB) has been used for analgesia of the thoracic wall since it was first described in 1905. A relatively recent alternative to the TPVB is the thoracic erector spinae plane (TESP) block, which involves the ultrasound-guided injection of local anesthetic into the interfascial plane deep to the erector spinae muscle at the level of the transverse process. It results in a loss of somatic sensory sensation across multiple unilateral dermatomes due to local anesthetic mediated blockade of the dorsal and ventral rami of the spinal nerve roots. It is increasingly being used due to ease of placing the block and a perception of greater safety. It has been shown to provide pain relief from rib fractures, thoracotomy, and chronic neuropathic pain of the chest wall. However, to date, TESP block has not been compared with TPVB in regards to analgesia with mastectomy surgery, which has been extensively studied.

The investigators hypothesize that TESP block will provide similar (i.e., non-inferior) analgesia compared to TPVB block while reducing the cumulative consumption of oral morphine equivalents during the 24h post-operative period. The two co-primary aims of the study are to compare a) pain scores at 2h post-operative period, and b) cumulative consumption of oral morphine equivalents during the 24h post-operative period. Secondary objectives include comparison between the group in terms of pain scores at 6, 12, 24, and 48 hours post-operatively, as well as block-related morbidity (e.g.- pneumothorax), time to perform each block, and opioid-related adverse effects (e.g.- postoperative nausea and vomiting).

ELIGIBILITY:
Criteria for Inclusion of Subjects:

* Female and male ASA physical status 1-3 scheduled for unilateral total mastectomy without immediate reconstruction
* Age 18-80 years old
* Able to participate personally or by legal representative in informed consent in English or Spanish

Criteria for Exclusion of Subjects:

* History of relevant drug allergy
* Age less than 18 or greater than 80 years
* Chronic opioid use or drug abuse
* Significant psychiatric disturbance
* Inability to understand the study protocol
* Refusal to provide written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Pain | 2 hours after surgery
  Pain score via Numeric Rating Scale (0-10)
Opioid Use | 24 hours after surgery
  Cumulative opioid consumption in oral morphine equivalents (mg)

SECONDARY OUTCOMES:
Pain | 6, 12, 24, and 48 hours after surgery
  Pain scores via Numeric Rating Scale (0-10)
Opioid morbidity | 2, 6, 12, 24, and 48 hours after surgery
  Any evidence of opioid-related morbidity or adverse effects
Procedural morbidity | 2, 6, 12, 24, and 48 hours after surgery
  Any evidence of procedure-related morbidity (i.e.- with paravertebral block and erector spinae plane block)
Time | preoperative
  Total time (in minutes) needed to perform the block (paravertebral or erector spinae plane block)

CONTACTS AND LOCATIONS:
Overall Officials: John C Alexander, MD, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No